CLINICAL TRIAL: NCT02149030
Title: Effectiveness of Cervical Screening in HPV Vaccinated Women - a Randomized Trial
Brief Title: Effectiveness of Cervical Screening in HPV Vaccinated Women
Acronym: HPV-004
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: European Union (Other); Academy of Finland (Other); Cancer Society of Finland (Unknown)
Responsible Party: Principal Investigator, Matti Lehtinen, Professor, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HPV-004
Record Dates: First submitted 2014-05-19; First posted 2014-05-29 (Estimated); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2/3

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- A1 (Active Comparator): A1) Cytological screening in A1 and A3. Frequent information of screening results for cytology and/or HPV DNA at the ages of 22 (cytology only), 25 and 30.
  Interventions: Other: Cytological screening in A1 and A3
- A2 (No Intervention): A2) infrequent information of screening results, only at the age 30 years.
- A3 (Other): A3) Cytological screening in A1 and A3. With at least 1000 participants is enrolled for interim safety analysis when the 1992 birth cohort is 25 years of age and cytology results are being revealed.
  Interventions: Other: Cytological screening in A1 and A3

INTERVENTIONS:
Other: Cytological screening in A1 and A3 — Cytological screening.
  Arms: A1; A3

SUMMARY:
The main objective of the study is to identify whether or not being informed infrequently results about screening is: 1) At least as safe and accurate as frequently obtaining all information from the present combination of opportunistic/organized cervical screening by comparing regimen results of three screening visits at the ages of 22, 25 and 30 years (Arm A1) vs. results of one screening visit at the age of 30 years (Arm A2) in Human papillomavirus (HPV) vaccinated young women.

DETAILED DESCRIPTION:
Altogether 16.500 1992-1995 born women vaccinated with the bi-valent human papillomavirus type 16 and 18 (HPV16/18) vaccine as adolescents either at the age of 12 to 15 or at the age of 18 will be invited to an effectiveness trial at the age of 22 years, and randomized into Arms A1 and A2, and A3, respectively.

Cervical samples and cervico-vaginal self-samples rinsed in first-void urine will be analysed for HPV and C. trachomatis DNA with MGP primer system followed by MALDITOF mass spectrometry on the SEQUENOM platform (HPV) and the Abbott™ PCR (Chlamydia trachomatis), respectively.

With assumed >50% participation the trial has 80% power to show non-inferiority of the infrequent vs. the frequent screening information.

A one-way (participant) blinded interim analysis among the 1992-born study participants in A1 and A3 arms, who have attended the 2nd study visit at the age of 25 years, will be performed in 2017 for assuring no statistically significant differences in the cervical intraepithelial neoplasia grade 2/3 (CIN2/CIN3) incidences of the two arms.

At the study end testing the null hypotheses of no difference in the incidence of the CIN2/3 end-points between the A1 and A2 intervention arms will be done using the Mantel-Haenszel one degree of freedom chi-square statistics.

ELIGIBILITY:
Inclusion Criteria:

* HPV 16/18 vaccinated. Born 1992-1995.

Exclusion Criteria:

* Immunocompromising disease. HPV 6/11/16/18 vaccination.

Ages: 22 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6958 (Actual)
Dates: Start 2014-03; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of intraepithelial neoplasia grade 2/3 (CIN2/3). | 2017-2020, i.e. four years (interim), 2021-2025, i.e. five years (final analysis). Participants will be followed for the duration of the study until 2026, an expected average of 9 years.
  1a) No marked difference in the incidence of CIN2/3 between arms A1 (participants frequently informed of the cytological results) and A3 (participants not informed of the cytological findings at the age of 22) (interim analysis). 1b) No difference in the incidence of CIN2/3 between arms A1 (participants frequently informed of the cytological results) and A2 (participants infrequently informed of the cytological results).
  The participants will be followed for 9 years starting from the year they turn 22. For 1992 born the follow-up will start in 2014 and end in 2023. For 1995 born the follow-up will start in 2017 and end in 2026.
  The interim analysis will include only 1992 cohort. The final analysis will include all cohorts (1992, 1993, 1994, 1995).

SECONDARY OUTCOMES:
Type-replacement | 2021-2025, i.e. four years
  Whether the post-vaccination distributions of vaccine-covered and/or non-vaccine covered HPV types develop differentially in the different vaccination arms by vaccination arm over time up to 15 years post vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Matti Lehtinen, MD, PhD, Principal Investigator — Tampere University
Locations (31):
- Finland (31):
  - Nuorisotutkimusasema: Tampereen yliopisto, Äänekoski
  - Nuorisotutkimusasema: Tampereen yliopisto, Hämeenlinna
  - HUS, Helsinki
  - Nuorisotutkimusasema: Tampereen yliopisto, Hyvinkää
  - Nuorisotutkimusasema: Tampereen yliopisto, Iisalmi
  - Nuorisotutkimusasema: Tampereen yliopisto, Jämsä
  - Nuorisotutkimusasema: Tampereen yliopisto, Joensuu
  - Nuorisotutkimusasema: Tampereen yliopisto, Jyväskylä
  - Nuorisotutkimusasema: Tampereen yliopisto, Kajaani
  - Nuorisotutkimusasema: Tampereen yliopisto, Kemi
  - Nuorisotutkimusasema: Tampereen yliopisto, Kokkola
  - Nuorisotutkimusasema: Tampereen yliopisto, Kotka
  - Nuorisotutkimusasema: Tampereen yliopisto, Kouvola
  - Nuorisotutkimusasema: Tampereen yliopisto, Kuopio
  - Nuorisotutkimusasema: Tampereen yliopisto, Lahti
  - Nuorisotutkimusasema: Tampereen yliopisto, Lappeenranta
  - Nuorisotutkimusasema: Tampereen yliopisto, Lohja
  - Nuorisotutkimusasema: Tampereen yliopisto, Mikkeli
  - THL, Oulu
  - Nuorisotutkimusasema: Tampereen yliopisto, Pori
  - Nuorisotutkimusasema: Tampereen yliopisto, Porvoo
  - Nuorisotutkimusasema: Tampereen yliopisto, Rauma
  - Nuorisotutkimusasema: Tampereen yliopisto, Rovaniemi
  - Nuorisotutkimusasema: Tampereen yliopisto, Salo
  - Nuorisotutkimusasema: Tampereen yliopisto, Savonlinna
  - Nuorisotutkimusasema: Tampereen yliopisto, Seinäjoki
  - Nuorisotutkimusasema: Tampereen yliopisto, Tampere
  - Nuorisotutkimusasema: Tampereen yliopisto, Turku
  - Nuorisotutkimusasema: Tampereen yliopisto, Vaasa
  - Nuorisotutkimusasema: Tampereen yliopisto, Vammala
  - Nuorisotutkimusasema: Tampereen yliopisto, Varkaus

REFERENCES:
- [Background] Vanska S, Luostarinen T, Baussano I, Apter D, Eriksson T, Natunen K, Nieminen P, Paavonen J, Pimenoff VN, Pukkala E, Soderlund-Strand A, Dubin G, Garnett G, Dillner J, Lehtinen M. Vaccination With Moderate Coverage Eradicates Oncogenic Human Papillomaviruses If a Gender-Neutral Strategy Is Applied. J Infect Dis. 2020 Aug 17;222(6):948-956. doi: 10.1093/infdis/jiaa099. PMID 32161969
- [Background] Louvanto K, Eriksson T, Gray P, Apter D, Baussano I, Bly A, Harjula K, Heikkila K, Hokkanen M, Huhtinen L, Ikonen M, Karttunen H, Nummela M, Soderlund-Strand A, Veivo U, Dillner J, Elfstom M, Nieminen P, Lehtinen M. Baseline findings and safety of infrequent vs. frequent screening of human papillomavirus vaccinated women. Int J Cancer. 2020 Jul 15;147(2):440-447. doi: 10.1002/ijc.32802. Epub 2019 Dec 16. PMID 31749143
- [Background] Gray P, Kann H, Pimenoff VN, Eriksson T, Luostarinen T, Vanska S, Surcel HM, Faust H, Dillner J, Lehtinen M. Human papillomavirus seroprevalence in pregnant women following gender-neutral and girls-only vaccination programs in Finland: A cross-sectional cohort analysis following a cluster randomized trial. PLoS Med. 2021 Jun 7;18(6):e1003588. doi: 10.1371/journal.pmed.1003588. eCollection 2021 Jun. PMID 34097688
- [Background] Kalliala I, Eriksson T, Aro K, Hokkanen M, Lehtinen M, Gissler M, Nieminen P. Preterm birth rate after bivalent HPV vaccination: Registry-based follow-up of a randomized clinical trial. Prev Med. 2021 May;146:106473. doi: 10.1016/j.ypmed.2021.106473. Epub 2021 Feb 24. PMID 33639181
- [Background] Lehtinen M, Gray P, Louvanto K, Vanska S. In 30 years, gender-neutral vaccination eradicates oncogenic human papillomavirus (HPV) types while screening eliminates HPV-associated cancers. Expert Rev Vaccines. 2022 Jun;21(6):735-738. doi: 10.1080/14760584.2022.2064279. Epub 2022 Apr 15. No abstract available. PMID 35404177
- [Background] Lehtinen M, Pimenoff VN, Nedjai B, Louvanto K, Verhoef L, Heideman DAM, El-Zein M, Widschwendter M, Dillner J. Assessing the risk of cervical neoplasia in the post-HPV vaccination era. Int J Cancer. 2023 Mar 15;152(6):1060-1068. doi: 10.1002/ijc.34286. Epub 2022 Oct 10. PMID 36093582
- [Background] Pimenoff VN, Gray P, Louvanto K, Eriksson T, Lagheden C, Soderlund-Strand A, Dillner J, Lehtinen M. Ecological diversity profiles of non-vaccine-targeted HPVs after gender-based community vaccination efforts. Cell Host Microbe. 2023 Nov 8;31(11):1921-1929.e3. doi: 10.1016/j.chom.2023.10.001. PMID 37944494
- [Background] Lehtinen M, Bruni L, Elfstrom M, Gray P, Logel M, Mariz FC, Baussano I, Vanska S, Franco EL, Dillner J. Scientific approaches toward improving cervical cancer elimination strategies. Int J Cancer. 2024 May 1;154(9):1537-1548. doi: 10.1002/ijc.34839. Epub 2024 Jan 9. PMID 38196123
- [Background] Lehtinen M, Elfstrom M, Vanska S, Dillner J. Elimination of cervical cancer by refined vaccination and screening. Int J Cancer. 2025 Feb 15;156(4):886-888. doi: 10.1002/ijc.35228. Epub 2024 Oct 25. No abstract available. PMID 39450703
- [Background] Louvanto K, Verhoef L, Pimenoff V, Eriksson T, Leppala S, Lagheden C, Gray P, Scibior-Bentkowska D, Sumiec E, Nieminen P, Dillner J, Berkhof J, Meijer CJLM, Lehtinen M, Nedjai B, Heideman DAM. Low methylation marker levels among human papillomavirus-vaccinated women with cervical high-grade squamous intraepithelial lesions. Int J Cancer. 2024 Nov 1;155(9):1549-1557. doi: 10.1002/ijc.35044. Epub 2024 May 27. PMID 38801336
- [Background] Taavela K, Eriksson T, Huhtala H, Bly A, Harjula K, Heikkila K, Hokkanen M, Nummela M, Kotaniemi-Talonen L, Lehtinen M, Louvanto K. The quality of life of frequently vs. infrequently screened HPV vaccinated women. Qual Life Res. 2024 Apr;33(4):941-949. doi: 10.1007/s11136-023-03575-y. Epub 2024 Jan 18. PMID 38238599
- [Background] Lehtinen M, Apter D, Baussano I, Eriksson T, Natunen K, Paavonen J, Vanska S, Bi D, David MP, Datta S, Struyf F, Jenkins D, Pukkala E, Garnett G, Dubin G. Characteristics of a cluster-randomized phase IV human papillomavirus vaccination effectiveness trial. Vaccine. 2015 Mar 3;33(10):1284-90. doi: 10.1016/j.vaccine.2014.12.019. Epub 2015 Jan 12. PMID 25593103